CLINICAL TRIAL: NCT05306418
Title: Safety, Efficacy and Exposure of Subcutaneously Administered NNC0365-3769 (Mim8) Prophylaxis in Children With Haemophilia A With or Without FVIII Inhibitors
Brief Title: A Research Study Looking at Mim8 in Children With Haemophilia A With or Without Inhibitors
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NN7769-4516; U1111-1255-1540 (Other: World Health Organization (WHO); 2020-003467-26 (EudraCT Number); jRCT2031220670 (Registry Identifier: jRCT)
Record Dates: First submitted 2022-03-23; First posted 2022-04-01 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Haemophilia A With or Without Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mim8 (Experimental): 52-week treatment period with a part 1 and part 2, where all participants receive Mim8 prophylaxis
  Interventions: Drug: Mim8

INTERVENTIONS:
Drug: Mim8 — For treatment part 1, all participants will start on once-weekly treatment and continue on this regimen until week 26. For treatment part 2, starting at week 26, all participants will be offered the choice to remain on once-weekly or switch to once-monthly dosing.
  Mim8 will be injected with a thin needle into the skin

SUMMARY:
This study is looking at how Mim8 works compared to other medicines in children with haemophilia A, who either have inhibitors or do not have inhibitors.

Mim8 is a new medicine that will be used for prevention of bleeds. Mim8 will be injected with a thin needle into the skin. The study will last for about 54-98 weeks, from screening to follow-up visit, In case the participant experiences bleeds, these can be treated with additional haemostatic medicine as agreed with the study doctor.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent obtained before any study-related activities. Study-related activities are any procedures that are carried out as part of the study, including activities to determine suitability for the study.
2. Male and female participants with the diagnosis of congenital haemophilia A of any severity based on medical records.
3. Aged 1-11 years (both inclusive) at the time of signing informed consent.
4. For previously treated participants :

   1. Participant has been prescribed treatment with FVIII concentrate or bypassing agent in the last 26 weeks prior to screening.
   2. Participants with endogenous FVIII activity greater than or equal to 1%, based on medical records, must have at least 1 treated bleed during the previous 26 weeks before screening for which factor VIII concentrate or bypassing agent has been prescribed (no requirements for participants with FVIII activity below 1%).
5. For previously untreated participants:

   a. Diagnosis of severe haemophilia A (endogenous FVIII activity below 1%) based on medical records.
6. Child and parent/caregiver willingness and ability to comply with scheduled visits and study procedures, including the completion of diary and patient-reported outcomes questionnaires.( For China mainland; assessed at the investigator's discretion unless otherwise stated.)

Exclusion criteria:

1. Known or suspected hypersensitivity to trial product or related products.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
2. Previous participation in this study. Participation is defined as signed informed consent.
3. Participation (i.e., signed informed consent) in any interventional clinical study with receipt of last dose within 6 months (or 5 half-lives of the investigational medicinal product, whichever is shorter) before planned randomisation.
4. Exposure to non-factor haemostatic products for bleeding prophylaxis within 6 months (or 5 half-lives of the medicinal product, whichever is shorter) before planned randomisation, for participants not included in the run-in.
5. Known congenital or acquired coagulation disorders other than haemophilia A.
6. Other conditions (e.g. autoimmune disease) or laboratory abnormality that may increase risk of bleeding or thrombosis, as evaluated by the investigator.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
7. Any disorder, except for conditions associated with haemophilia A, that in the investigator's opinion might jeopardise the participant's safety or compliance with the protocol.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
8. Mental incapacity, unwillingness to cooperate or a language barrier precluding adequate understanding and cooperation.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
9. Lack of adequate parental/caregiver support to enter accurately and timely information regarding treatment and bleeding episodes into an (electronic) diary.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
10. Previous or current treatment for thromboembolic disease (with the exception of previous catheter-associated thrombosis for which anti-thrombotic treatment is not currently ongoing) or signs of thromboembolic disease.
11. Major surgery planned to take place after screening.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
12. Immune tolerance induction planned to take place after treatment initiation.(For China mainland; assessed at the investigator's discretion unless otherwise stated.)
13. Hepatic dysfunction defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) greater than 3 times the upper limit of normal combined with total bilirubin greater than 1.5 times the upper limit of normal measured at screening.
14. Serum creatinine above 1.5 x upper limit of normal (ULN), measured at screening.
15. Pregnancy (female participants).(Will be assessed at investigator's discretion, according to suspicion of pregnancy.)

Ages: 1 Year to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-11-13 (Actual); Study Completion 2024-11-13 (Actual)

PRIMARY OUTCOMES:
Number of treatment emergent adverse events | From treatment initiation to follow up visit (week 0 to week 72)
  Count of events

SECONDARY OUTCOMES:
Number of treated bleeds | From treatment initiation to end of treatment (week 0 to week 52)
  Count of bleeds
Number of treated spontaneous bleeds | From treatment initiation to end of treatment (week 0 to week 52)
  Count of bleeds
Number of treated traumatic bleeds | From treatment initiation to end of treatment (week 0 to week 52)
  Count of bleeds
Number of treated joint bleeds | From treatment initiation to end of treatment (week 0 to week 52)
  Count of bleeds
Number of treated target joint bleeds | From treatment initiation to end of treatment (week 0 to week 52)
  Count of bleeds
Number of injection site reactions | From treatment initiation to end of treatment (week 0 to week 52)
  Count of reactions
Consumption of factor product per bleed treatment (number of injections) | From run-in initiation to end of treatment (week -26 to week 52)
  Count of injections
Occurrence of anti-Mim8 antibodies | From treatment initiation to end of treatment (week 0 to week 52)
  Count of participants
Mim8 plasma concentration | From treatment initiation to end of treatment (week 0 to week 52)
  µg/mL
Change in physical function domain of PEDS QL (Paediatric Quality of Life inventory) Generic Core Scales | From treatment initiation to end of treatment (week 0 to week 52)
  Score on a scale 0-100 (applies for scale scores and total score). A higher score indicates a better health-related quality of life
Treatment preference for Mim8 versus previous treatment using Caregiver H PPQ (Caregiver Haemophilia Patient Preference ) | Once during treatment (week 26)
  Percentage of participants
Change in participants' treatment burden using the Hemo TEM (Haemophilia treatment experience measure) | From treatment initiation to end of treatment (week 0 to week 52)
  Score on a scale 0-100 (applies for scale scores and total score). A lower score indicates a lower treatment burden.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (52):
- United States (9):
  - Children's Hospital Los Angeles - Endocrinology, Los Angeles, California
  - Univ of Colorado Sch of Med, Aurora, Colorado
  - St Joseph's Hospital Foundation, Tampa, Florida
  - Children's Healthcare Atlanta, Atlanta, Georgia
  - Children's Hospital at Memorial Health, Savannah, Georgia
  - University of Iowa_Iowa City, Iowa City, Iowa
  - Univ Hosp Cleveland Med Ctr, Cleveland, Ohio
  - Penn State MS Hershey Med Ctr, Hershey, Pennsylvania
  - St Christopher Hosp for Child, Philadelphia, Pennsylvania
- Canada (2):
  - McMaster Children's Hospital, Hamilton, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
- China (6):
  - Beijing Children's Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Children's Hospital，Capital Medical University, Beijing, Beijing Municipality
  - Nanfang Hospital, Southern Medical University-Haematology, Guangzhou, Guangdong
  - Chengdu Women's and Children's Central Hospital, Chengdu, Sichuan
  - Institute of Hematology and Blood Diseases Hospital, Tianjin-Hematology, Tianjin, Tianjin Municipality
  - Children's Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
- Universitätsklinikum Bonn - Institut für Experimentelle Hämatologie, Bonn, Germany
- India (5):
  - Nirmal Hospital Pvt. Ltd., Surat, Gujarat
  - Seth GS Medical College & KEM Hospital, Mumbai, Maharashtra
  - Sahyadri Super Speciality Hospital, Pune, Maharashtra
  - J K Lon Hospital, Jaipur, Rajasthan
  - Post Graduate Institute of Child Health, Noida, Uttar Pradesh
- Sheba MC - The Israeli National Hemophilia Center, Tel Litwinsky, Israel
- Italy (2):
  - Ospedale Pediatrico Bambino Ges, Rome
  - A.O.U. Città della Salute e della Scienza di Torino-Ospedale, Torino
- Japan (4):
  - Ota Memorial Hospital_Pediatrics, Gunma
  - Sapporo Tokushukai Hospital_Pediatrics, Hokkaido
  - Saitama Children's Med Centre_Hematology-Oncology, Saitama
  - Ogikubo Hospital_Pediatries & Blood, Tokyo
- Children Oncohaematology department Children's Hospital,, Vilnius, Lithuania
- Netherlands (2):
  - Academisch Medisch Centrum, Amsterdam
  - UMC Utrecht, Van Creveldkliniek, Utrecht
- Poland (3):
  - Uniwersytecki Szpital Kliniczny im. J.Mikulicza-Radeckiego, Wroclaw, Lower Silesian Voivodeship
  - CSK UM Uniwersyteckie Centrum Pediatrii im. M. Konopnickiej, Lodz
  - Uniwersytecki Szpital Dzieciecy, Dzial Krwiolecznictwa, Lublin
- Portugal (2):
  - Unidade Local de Saúde São José EPE- Hospital D. Estefânia, Lisbon
  - ULS São João, E.P.E., Porto
- Russia (4):
  - SAHI Kuzbass Hospital(former Regional clinical hospital), Kemerovo
  - Children Regional Clinical Hospital, Krasnodar
  - Morozovskaya municipal children hospital, Moscow
  - Republican Hospital n.a. V. A. Baranov, Petrozavodsk
- Charlotte Maxeke Johannesburg Academic Hospital, Parktown, Johannesburg, Gauteng, South Africa
- South Korea (2):
  - Daejeon Eulji Medical Center, Eulji University, Daejeon
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (2):
  - Hospital Sant Joan de Déu, Esplugues Llobregat
  - Hospital Universitario La Paz, Madrid
- Switzerland (2):
  - Universitätsklinik für Kinderheilkunde, Bern
  - Pädiatrische Onkologie-Hämatologie, Lucerne
- National Taiwan University Children's Hospital, Taipei, Taiwan
- United Kingdom (2):
  - Arthur Bloom Haemophilia Centre, Cardiff
  - St Thomas' Hospital - Haemostasis and Thrombosis Centre, London

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com